CLINICAL TRIAL: NCT00790660
Title: A Phase 2a, Randomized, Double-Blind, Placebo Controlled, Multiple Dose Study to Assess the Safety and Tolerability of ASP1941 in Adult Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Assess the Safety and Tolerability of ASP1941 in Adults With Type 2 Diabetes Mellitus.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1941-CL-0016
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: ASP1941; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ipragliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- ASP1941 Lowest Dose (Experimental): Oral
  Interventions: Drug: ASP1941
- ASP1941 Low Dose (Experimental): Oral
  Interventions: Drug: ASP1941
- ASP1941 Medium Dose (Experimental): Oral
  Interventions: Drug: ASP1941
- ASP1941 High Dose (Experimental): Oral
  Interventions: Drug: ASP1941
- Placebo (Placebo Comparator): Oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP1941 — Oral
  Arms: ASP1941 High Dose; ASP1941 Low Dose; ASP1941 Lowest Dose; ASP1941 Medium Dose
Drug: Placebo — Oral
  Arms: Placebo

SUMMARY:
This study is intended to assess safety and tolerability of ASP1941 compared to placebo in adult subjects with type 2 diabetes mellitus

DETAILED DESCRIPTION:
Trial includes a two week washout period before entering the treatment period for subjects on oral anti-diabetic medication.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of type 2 diabetes mellitus
* HbA1c value between 7.0 and 10.0%
* Body mass index between 20 and 45 kg/m2

Exclusion Criteria:

* Established diagnosis of type 1 diabetes mellitus
* Serum creatinine > upper limit of normal range
* Proteinuria (microalbumin/creatinine ratio > 300 mg/g)
* Urinary tract infection
* Severe uncontrolled Hypertension
* Significant renal, hepatic or cardiovascular disease
* HIV Positive
* History of drug or alcohol abuse/dependency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-10-23 (Actual); Primary Completion 2009-03-06 (Actual); Study Completion 2009-03-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety through clinical safety labs and adverse events | 6 Weeks

SECONDARY OUTCOMES:
Evaluation of routine PK and PD parameters | 6 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: use Central Contact, Study Director — Astellas Pharma Global Development
Locations (1):
- San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/study.aspx?ID=3